CLINICAL TRIAL: NCT01439984
Title: A Randomized, Double-blind, Placebo-controlled, Fixed Dose, Parallel Grouped, Multi-center Clinical Study to Evaluate the Safety and Efficacy of PED-1 in Male Patients With Premature Ejaculation
Brief Title: Trial of PED-1 in Male Patients With Premature Ejaculation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Symyoo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTC-PE-01
Record Dates: First submitted 2011-09-18; First posted 2011-09-23 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-10

CONDITIONS: Premature Ejaculation
Keywords: PE; IELT; DCIT
MeSH Terms: conditions — Premature Ejaculation | interventions — Clomipramine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PED-1 (Experimental): PED-1 (Clomipramine 15 mg)
  Interventions: Drug: Clomipramine
- placebo (Placebo Comparator)
  Interventions: Drug: Clomipramine

INTERVENTIONS:
Drug: Clomipramine — Clomipramine 15 mg tablet or placebo tablet on demand for 12 weeks
  Other Names: PED-1

SUMMARY:
The purpose of this study is to evaluate whether PED-1 is more effective than Placebo in the treatment of premature ejaculation.

DETAILED DESCRIPTION:
This study is to evaluate whether PED-1 is effective than Placebo in the treatment of premature ejaculation. The patients will be randomized and allocated to two treatment groups into placebo, PED-1. The criteria for Intravaginal Ejaculation Latency Time(IELT) for enrollment will be > or =2 min in the at least 75% of the sexual intercourse. To diagnosis premature ejaculation, the PEDT(Premature Ejaculation Diagnosis Tool) will be used. The patients undergone drug free baseline period will take test drugs for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent for subjects and partners
* Men 20-65 ages
* Stable monogamous relation at least for 6 mo
* Premature Ejaculation Diagnosis Tool (PEDT) more than 9
* At least 6 mo of premature ejaculation Hx
* IELT of =< 2 min in >= 75% of evaluable events during 4 week screening period

Exclusion Criteria:

* History of medical or psychiatric illness
* Erectile dysfunction (<21 International Index of Erectile Function-Erectile Function (IIEF-EF) domain score) or other forms of sexual dysfunction
* Partner sexual dysfunction
* Known hypersensitivity to clomipramine and contraindications for clomipramine

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2011-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Intravaginal ejaculation latency time (IELT)(seconds) | 12 weeks

SECONDARY OUTCOMES:
Drug coitus interval time (hours) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Whan-Seok Choi, MD,PhD, Principal Investigator — Seoul St. Marry's Hospital
Locations (5):
- South Korea (5):
  - Inje University Ilsan Paik Hospital, Goyang-si, Gyeonggi-do
  - National Health Insurance Corporation Ilsan Hospital, Goyang-si, Gyeonggi-do
  - Uijeongbu St.Marry's Hospital, Uijeongbu-si, Gyeonggi-do
  - Ewha Womans University Mokdong Hospital, Seoul
  - Seoul St.Marry's Hospital, Seoul